CLINICAL TRIAL: NCT05759494
Title: The Clinical and Pharmacoeconomic Impact of Rapid Diagnostic Test (Multiplex PCR FilmArray) on Antimicrobial Decision Making Compared to Conventional Decision Making Among Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Fakher, assistant professor, Cairo University
Other Study IDs: MD-37-2022
Record Dates: First submitted 2022-09-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: 50 patients before use rapid diagnostic test (multiplex PCR filmArray)
- B: 50 patients after use rapid diagnostic test (multiplex PCR filmArray)
  Interventions: Diagnostic Test: rapid diagnostic test (multiplex PCR filmArray)

INTERVENTIONS:
Diagnostic Test: rapid diagnostic test (multiplex PCR filmArray) — novel diagnostic platform, the "FilmArray®", which combines automated sample preparation, nucleic acid extraction and PCR-based detection of 31 separate targets from a single unprocessed sample in one hour. It combines nesting and multiplexing of the PCR (referred to here as nested multiplex or "nmPCR") together with DNA melting curve analysis.
  Groups: B

SUMMARY:
We will show in this study the impact of use the rapid diagnostic method (multiplex PCR filmArray) on clinical and pharmacoeconomic aspects among Critically Ill Patients.

DETAILED DESCRIPTION:
Prospective and retrospective study on 100 patients complaining from sepsis in intensive care unit in International Medical center. Two phase study 50 patients before and 50 patients after use rapid diagnostic test (multiplex PCR filmArray)

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Critically ill patients admitted to ICU, diagnosed as sepsis.

Exclusion Criteria:

* Surviving time less than 48 hours.

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 male and female patients, age between 16 and 85. One-year study 6 months before and 6 months after using the rapid diagnostic test.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
clinical | through study completion, an average of 1 year
  Clinical resolution of sepsis ( by percentage)
Pharmacoeconomic | through study completion, an average of 1 year
  1-Reduction of cost and reduction of respective antimicrobial cases (by percentage )
clinical | through study completion, an average of 1 year
  survival (by percentage )
clinical | through study completion, an average of 1 year
  length of stay in ICU (by days)
clinical | through study completion, an average of 1 year
  change strategy of antibiotic in first week (by percentage)
pharmacoeconomic | through study completion, an average of 1 year
  DOT of antimicrobial (by days )

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018 Jun;44(6):925-928. doi: 10.1007/s00134-018-5085-0. Epub 2018 Apr 19. No abstract available. PMID 29675566
- [Result] Peeters P, Ryan K, Karve S, Potter D, Baelen E, Rojas-Farreras S, Rodriguez-Bano J. The impact of initial antibiotic treatment failure: real-world insights in patients with complicated, health care-associated intra-abdominal infection. Infect Drug Resist. 2019 Jan 31;12:329-343. doi: 10.2147/IDR.S184116. eCollection 2019. PMID 30774399
- [Result] Poritz MA, Blaschke AJ, Byington CL, Allen L, Nilsson K, Jones DE, Thatcher SA, Robbins T, Lingenfelter B, Amiott E, Herbener A, Daly J, Dobrowolski SF, Teng DH, Ririe KM. FilmArray, an automated nested multiplex PCR system for multi-pathogen detection: development and application to respiratory tract infection. PLoS One. 2011;6(10):e26047. doi: 10.1371/journal.pone.0026047. Epub 2011 Oct 19. PMID 22039434
- See also: Definitions of sepsis and septic shock were last revised in 2001. Considerable advances have since been made into the pathobiology (changes in organ function, morphology, cell biology, biochemistry, immunology, and circulation), management, and epidemiol — https://pubmed.ncbi.nlm.nih.gov/26903338/
- See also: he antibiotic use and resistance can contribute to the rates of sepsis hospitalization and mortality — https://pubmed.ncbi.nlm.nih.gov/29675566/
- See also: However, approximately 20-30% of initial antibiotic treatment was reported to be ineffective in patients. Thus, further delay of effective antibiotic treatment could increase the risk of mortality — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6362915/
- See also: Here we use a novel diagnostic platform, the "FilmArray®", which combines automated sample preparation, nucleic acid extraction and PCR-based detection of 31 separate targets from a single unprocessed sample in one hour. — https://pubmed.ncbi.nlm.nih.gov/22039434/